CLINICAL TRIAL: NCT05194657
Title: Assessment of Reading Performance in Patients With Acrysof IQ Vivity Toric or Non-toric vs Monofocal Acrysof IQ Toric or Non-toric IOL
Brief Title: Reading Performance in Patients With Acrysof IQ Vivity Versus Acrysof IQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vivity
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Cataract
Keywords: Cataract; Cataract surgery; ehanced depth of focus intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acrysof IQ Vivity (Experimental): Patient will receive the enhanced depth of focus IOL during cataract surgery
  Interventions: Device: enhanced depth of focus IOL
- Acrysof IQ (Experimental): Patiet will receive the monofocal IOL during cataract surgery
  Interventions: Device: monofocal IOL

INTERVENTIONS:
Device: enhanced depth of focus IOL — Acrysof IQ Vivity, enhanced depth of focus IOL
  Arms: Acrysof IQ Vivity
Device: monofocal IOL — Acrysof IQ, monofocal IOL
  Arms: Acrysof IQ

SUMMARY:
Comparison of the visual function and reading performance between the Acrysof IQ Vivity IOL, an EDOF IOL, and the monofocal Acrysof IQ.

DETAILED DESCRIPTION:
With increasing demands of patients concerning their visual function after cataract surgery, a variety of advanced technology intraocular lenses (IOL) have become available in the last years. Various developments aim at a reduced spectacle independence for patients after cataract or refractive lens surgery.

Novel technology for providing an extended depth of focus (EDOF) has been developed to account for unmet needs of patients. A novel EDOF IOL, the Acrysof IQ Vivity, has two surface transition elements that work simultaneously by stretching and shifting the wavefront to create a continuous extended focal range instead of multiple focal points.

To assess the performance of such an IOL technology, most studies assess visual acuity at different distances from far, to intermediate up to near. Since most activites with digital devices implicate reading, it is not surprising that reading difficulty is the most common complaint among individuals experiencing visual disturbances with multifocal designs.

Reading ability is usually evaluated using various reading tests that assess reading speed and reading acuity defined as the print size that can stell be read with sufficient speed. However, one of the fundamental problems of these tests is that reading speed is also influenced by the average amount of time that a patient reads as well as the language of the text, whether it is the first or second language.

A novel method to analyse reading performance that appears to be more objective and less reliant on the cognitive abilities of the patient is the observation of the reading pattern using a high-speed eye-tracking system that analyses eye fixations during the reading test. In previous studies we have seen that several aspects of this reading patter, i.e. fixation duration and fixation frequency, appear to correlate with the reading performance overall and can be differentially used to discriminate between cognitive and visuo-motor processing.

Hence, the aim of this study is to assess the visual function and reading performance with an EDOF IOL (Acrysof IQ Vivity) compared to a standard monofocal IOL (Acrysof IQ).

136 eyes of 68 patients will be included into this study. According to the randomization, 34 patients will be implanted with the Acrysof IQ Vivity in both eyes and the other 34 patients will be implanted with the Acrysof IQ in both eyes. A follow-up examination will be performed at 3 months postoperative. During this visit a slitlamp examination, biometry and tomography of the eye, refraction and visual acuity assessment, an OCT examination, a retroillumination photogrypha, reading speed analysis and halometry will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Stereopsis
* age 21 and older
* regular corneal astigmatism of up to 3.0 D
* written informed consent prior to surgery
* normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* availability, willingness and sufficient cognitive awareness to comply with examination procedures
* german as mother-tongue
* calculated IOL power needed is below 15.0 D or above 25.0 D (no high myopia or high hypermetropia will be recruited)

Exclusion Criteria:

* relevant other ophthalmic diseases such as: pseudoexfoliation, glaucoma, traumatic cataract, corneal scars, and other co-morbidity that could affect capsule bag stability (e.g. Marfan syndrome) or retinal diseases affecting visual acuity (AMD, Macular Pucker, post-operative macular edema...)
* amblyopia
* contact lenses
* irregular corneal astigmatism on corneal topography
* postoperative subjective refraction smaller/ higher than or 0.75 D
* pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-01-03 (Estimated); Study Completion 2024-01-03 (Estimated)

PRIMARY OUTCOMES:
Reading speed | 24 months
  reading speed will be assessed with the Eyetracker device at 66 centimetres and will be compared between the EDOF IOL and the monofocal IOL

SECONDARY OUTCOMES:
Visual acuity | 24 months
  Visual acuity will be assessed using the ETDRS charts and will be compared between the EDOF IOLs and the monofocal IOLs

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amir-Asgari S, Georgiev S, Ruiss M, Plainis S, Pilwachs C, Findl O. Comparing postoperative reading performance and visual outcomes of a non-diffractive EDOF-IOL versus a monofocal IOL: a randomized controlled eye movement study. BMC Ophthalmol. 2025 Dec 24;25(1):694. doi: 10.1186/s12886-025-04507-9. PMID 41444551